CLINICAL TRIAL: NCT03729219
Title: A Randomized, Placebo-controlled Phase II b(OEV 123) Study to Evaluate Safety, Immunogenicity, Diagnostic Methodology, and Estimate Vaccine Efficacy of an Oral Enterotoxigenic Escherichia Coli(ETEC) Vaccine(ETVAX) for Prevention of Clinically Significant ETEC Diarrhea in Healthy Adult Travelers Visiting West Africa
Brief Title: Prevention of Diarrheal Disease Due to Infection With Enterotoxigenic E. Coli (ETEC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scandinavian Biopharma AB (Industry)
Collaborators: Göteborg University (Other); United Medix Laboratories Ltd. (Unknown); Oy Medfiles Ltd (Industry); University of Helsinki (Other); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OEV 123
Record Dates: First submitted 2017-10-16; First posted 2018-11-02 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled phase IIb
Who Masked: Participant, Care Provider, Investigator
Masking Description: Other parts will be blinded except unblinded person who prepares the doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETVAX (Experimental): Contains inactivated Tetravalent ETEC vaccine, 10 ug Double-mutant heat-labile toxin (dmLT) and effervescent power for oral solution administered twice 14 (plus minus 7) days intervals.
  Interventions: Biological: E. coli ETVAX
- Placebo (Placebo Comparator): Effervescent power for oral solution administered wice 14 (plus-minus 7) days intervals
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: E. coli ETVAX — Oral suspension Sterile water is added to dmLT . Vaccine is poured to the effervescent solution and needed amount of dmLT is added.
  Arms: ETVAX
Other: Placebo — Oral suspension
  Arms: Placebo

SUMMARY:
This is a Phase II b, double-blind, randomized, placebo-controlled study in healthy adults (age 18-65 years) to evaluate the safety, immunogenicity, different diagnostic tools and efficacy of ETVAX. Participants will travel to Grand Popo, Africa for 12 days. Prior travelling participants will be vaccinated with two doses of vaccine or placebo. Vaccine Preventable Outcome will be identified and then characterized as to incidence, duration, severity and frequency of Moderate or Severe Travellers diarrhea. Health related information and assessments will be recorded during the travel.

DETAILED DESCRIPTION:
This is a Phase II b, double-blind, randomized, placebo-controlled study in healthy adults (age 18-65 years) to evaluate the safety, immunogenicity, different diagnostic tools and efficacy of two doses of ETVAX. Study participants will be recruited among students, and personnel at the University of Helsinki and Helsinki University Hospital and among those responding to recruitment advertisements. To be eligible, the participants have to commit themselves to comply with the study protocol which involves in addition to vaccination, study visits and sampling, and commitment to travel to Grand Popo, Benin and stay there for 12 days. After providing written informed consent, eligible participants will be randomized (ratio 1:1, and block randomization in groups of 6) and immunized with two doses of vaccine or placebo, given 14±7 days apart while in Finland. The last dose of vaccine will be administered at least one week before departure (and no more than 30 days prior to travel) to Benin. Eligible participants will pay four pre-travel visits (V0 + V 1-3) to Aava Travel Clinic / University of Helsinki prior to travel. They will be asked to fill in pre-travel questionnaire latest at visit 1 (Q1) and fill in an Adverse Event Form (AEF1 and AEF2) after each dose, and give blood and fecal samples and saliva before travel. The participants will go together to Benin in groups of 25-35 individuals at a time.

In Benin, the participants will be seen within 48 hours of arrival to the study site in Grand Popo. Once the participants arrive at the study site in Grand Popo, they will be provided with practical information and contact details of the study personnel. They will receive the health card (HC1) and a stool collection kit with instructions.

Diarrhea reporting, stool collection, and stool submission procedures will be reviewed with the study participants. One routine visit at day 4 is planned for review of the participant's health status and collection of a routine stool sample. Other visits will take place when and if the participant gets Travelers Diarrhea (TD) episodes for collection of study specific stool samples and health related information and assessments. If more than one diarrhea episode occurs, 48 diarrhea and symptom (TD defined symptoms) free hours must have passed between the episodes for the new episode to be counted as a separate one. One or two days prior to departure from the Grand Popo site, all participants will have a final review of their HC1s. Health Card ( HC2) will be given. After 1-6 days back in Finland the participant has to give blood and a routine stool sample and they fill in Questionnaire 2 (Q2), HC2 will be reviewed. Approx. 30 days after return to Finland the last stool and blood sample will be collected and the post-travel questionnaire (Q3) filled and HC2 reviewed. Participants who get urinary tract infection will fill in Urinary questionnaire 4 (QU4) form at the time of infection. This follow-up is valid until V5.

ELIGIBILITY:
Inclusion criteria:

1. Male or female age ≥18 and ≤ 65 years
2. General good health at the time of first vaccination
3. Female participants of childbearing potential must not be pregnant
4. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study
5. Willingness to participate in the study after all aspects of the protocol have been explained and written informed consent obtained
6. Availability for the study duration, including all planned follow-up visits
7. Intake of atovaquone + proguanil (Malarone) as anti-malaria prophylax according to prescription guidelines mandatory before, during and after travel to Benin

Exclusion Criteria:

1. Presence of a significant medical or psychiatric condition, which in the opinion of the investigator precludes participation in the study
2. Known or suspected history of drug, chemical or alcohol abuse, as deemed by the investigator/physician; AUDIT > 13 points
3. Known recent history of impaired immune function which, according to the judgement of the investigator could influence the immune response
4. Intends to receive any other investigational vaccine during the study period, or within two weeks prior to study vaccination
5. Intends to donate blood at any time during the study.
6. An acute or chronic medical condition that, in the opinion of the investigator/physician, would render ingestion of the investigational products unsafe or would interfere with the evaluation of responses. This includes, but is not limited to gastrointestinal diseases and autoimmune diseases requiring treatment
7. Any history of psychosis or bipolar disorder or on-going significant mental disorder
8. Regular (daily) use of laxatives or agents which lower stomach acidity (antacids, proton pump inhibitors) less than one week before visit V1
9. Use of any oral or parenteral medication known to affect the immune function (e.g., corticosteroids and others) within 30 days preceding the first vaccination or planned use during the active study period
10. Traveled to ETEC-endemic areas within the last year or visit for > two months in ETEC endemic areas during the last 10 years
11. Receipt of Dukoral or other ETEC or cholera vaccines within 3 years or planned receipt of such vaccine except ETVAX during the study
12. Antibiotic therapy within two weeks prior to the vaccination
13. History of diarrhea in the 7 days prior to vaccination (defined as ≥ 3 unformed loose stools in 24 hours)
14. Any other criteria which, in the investigator's opinion, would compromise the ability of the traveler to participate in the study, the safety of the study, or the results of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Safety: Number of vaccine attributable adverse events | From first vaccination until leave for Benin, approximately 13-50 days
  Number of vaccine attributable adverse events
Immunogenicity: Fold change of serum titers of IgA and IgG against LTB | Change from baseline (just before first vaccination) to Visit 3 (5-6 days after second vaccination), an average of 20 days
  Fold change of serum titers of Immunoglobulin A (IgA) and Immunoglobulin G (IgG) against heat-labile toxin (LTB)
Immunogenicity: Number of subjects responding to heat-labile toxin (LTB) | Change from baseline (just before first vaccination) to Visit 3 (5-6 days after second vaccination), an average of 20 days
  Number of subjects responding to heat-labile toxin (LTB) based on serum Immunoglobulin A (IgA) and Immunoglobulin G (IgG) (i.e. fold change at least 2)
Immunogenicity: Fold change of serum titers of Immunoglobulin A (IgA) and Immunoglobulin G (IgG) against O78 lipopolysaccharide (LPS) | Change from baseline (just before first vaccination) to Visit 3 (5-6 days after second vaccination), an average of 20 days
  Fold change of serum titers of Immunoglobulin A (IgA) and Immunoglobulin G (IgG) against O78 lipopolysaccharide (LPS)
Immunogenicity: Number of subjects responding to O78 lipopolysaccharide (LPS) | Change from baseline (just before first vaccination) to Visit 3 (5-6 days after second vaccination), an average of 20 days
  Number of subjects responding to O78 lipopolysaccharide (LPS) based on serum Immunoglobulin A (IgA) and Immunoglobulin G (IgG) (i.e. fold change at least 2)
Diagnostic Tools:To set the optimal threshold limits of the two quantitativePolymerase chain reaction (PCR ) procedures | 12 days in Benin and 30 days post-travel in Finland, approximately 42 days
  To set the optimal threshold limits of the two quantitative Polymerase chain reaction (PCR ) procedures by setting limits for the number of amplification cycles (Cq values) which best allows (in terms of sensitivity, specificity, and positive predictive value) for identification of clinically significant ETEC TD cases, as well as cases associated with other enteric pathogens using the culture based bacterial detection method as the "Gold standard" for comparison.

SECONDARY OUTCOMES:
Efficacy: The incidence of Vaccine Preventable Outcomes (VPO) | 12 days in Benin and 30 days post-travel in Finland, approximately 42 days
  The incidence of cases with moderate or severe ETEC VPO diarrhea in the vaccinated and placebo groups of travelers.
Diagnostic Tools:Extent to which the non-culture based PCR assays can help resolve mixed ETEC infections | 12 days in Benin and 30 days post-travel in Finland, approximately 42 days
  Percentage of clinically significant Traveller's Diarrhea cases with mixed infection where decision about what is the primary causative agent is concordant between Amphidial qPCR method and culture-based antigen detection method
Diagnostic Tools:The extent to which the TaqMan array yields results for ETEC colonization factor that are comparable to those obtained by culture based methods. | 12 days in Benin and 30 days post-travel in Finland, approximately 42 days
  Percentage of clinically significant Traveller's Diarrhea cases with mixed infection where decision about what is the primary causative agent is concordant between TaqMan arrays qPCR method and culture-based antigen detection method

CONTACTS AND LOCATIONS:
Overall Officials: Anu Kantele, Principal Investigator — University of Helsinki, Dept. of Infectious Diseases
Locations (1):
- Lääkärikeskus Aava, matkailuklinikka, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu J, Jokiranta TS, Carlin N, Stroup S, Zhang J, Sjostrand B, Svennerholm A-M, Houpt ER, Kantele A. Use of a TaqMan Array Card for identification of enterotoxins and colonization factors directly from stool samples in an enterotoxigenic E. coli vaccine study. Microbiol Spectr. 2025 Mar 4;13(3):e0187024. doi: 10.1128/spectrum.01870-24. Epub 2025 Feb 11. PMID 39932427